CLINICAL TRIAL: NCT03326856
Title: Clinical Trial to Evaluate ET-01 in Subjects With Lateral Canthal Lines
Brief Title: ET-01 in Subjects With Lateral Canthal Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eirion Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ET-01-LCL-206
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Results first posted 2021-09-10 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Lateral Canthal Lines; Crow's Feet
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: sequential, dose escalating study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Vehicle (Placebo Comparator): Vehicle
  Interventions: Biological: Vehicle
- Dose 1 (Experimental): botulinum toxin, Type A, Dose 1
  Interventions: Biological: botulinum toxin, Type A
- Dose 2 (Experimental): botulinum toxin, Type A, Dose 2
  Interventions: Biological: botulinum toxin, Type A
- Dose 3 (Experimental): botulinum toxin, Type A, Dose 3
  Interventions: Biological: botulinum toxin, Type A
- Dose 4 (Experimental): botulinum toxin, Type A, Dose 4
  Interventions: Biological: botulinum toxin, Type A

INTERVENTIONS:
Biological: botulinum toxin, Type A — topical liniment
  Other Names: ET-01
  Arms: Dose 1; Dose 2; Dose 3; Dose 4
Biological: Vehicle — Vehicle Formulation
  Arms: Vehicle

SUMMARY:
This study tests an investigational drug formulation called ET-01, botulinum toxin, Type A, topical, in lateral canthal lines (LCL).

DETAILED DESCRIPTION:
This product is being tested for its ability to reduce lateral canthal lines, also known as Crow's Feet.

ELIGIBILITY:
Inclusion Criteria:

* 25 - 65 years of age
* minimal to moderate Crow's Feet wrinkles at rest
* moderate to severe Crow's Feet wrinkles on contraction
* willingness to refrain from any product affecting skin remodeling
* female subjects must be not pregnant and non-lactating-

Exclusion Criteria:

* history of adverse reactions to any prior botulinum toxin treatments
* history of vaccination or non-response to any prior botulinum toxin treatments
* botulinum toxin treatment in the prior 6 months
* present or history of neuromuscular disease, eyelid ptosis, muscle weakness, paralysis, or "dry eye"
* history of peri-ocular surgery, brow lift or related procedures
* procedures affecting the lateral canthal region in the prior 12 months
* application of topical prescription medication to the treatment area
* female subjects who are pregnant or are nursing a child

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Theobald, MD, PhD, Study Director — Eirion Therapeutics
Locations (1):
- Cary Skin Care, Cary, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose 1: botulinum toxin, Type A, topical liniment Dose 1x on Day 0
- Dose 2: botulinum toxin, Type A, topical liniment Dose 1.8x on Day 0
- Dose 3: botulinum toxin, Type A, topical liniment Dose 2.5x on Day 0
- Dose 4: botulinum toxin, Type A, topical liniment Dose 3.5x on Day 0
Period: Overall Study
Arm/Group | Vehicle | Dose 1 | Dose 2 | Dose 3 | Dose 4
Started | 13 | 9 | 9 | 9 | 8
Completed | 12 | 8 | 9 | 9 | 8
Not Completed | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Total
Number analyzed (Participants) | 13 | 9 | 9 | 9 | 8 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 9 | 9 | 9 | 8 | 48
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 9 | 7 | 8 | 43
  Male | 2 | 1 | 0 | 2 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 13 | 8 | 9 | 8 | 8 | 46
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 9 | 9 | 9 | 8 | 48
IGA-C [Mean (Standard Deviation); unit: units on a scale] — Investigator Global Assessment on Contraction using the ordinal Crow's Feet Wrinkle Scale where severity is scored between 0=absent and 4=severe.
  units on a scale | 3.5 (0.4) | 3.6 (0.5) | 3.4 (0.5) | 3.4 (0.5) | 3.5 (0.5) | 3.5 (0.5)
SSA-C [Mean (Standard Deviation); unit: units on a scale] — Subject Self-Assessment on Contraction using the ordinal Crow's Feet Wrinkle Scale where severity is scored between 0=absent and 4=severe.
  units on a scale | 3.5 (0.5) | 3.6 (0.5) | 3.4 (0.5) | 3.5 (0.5) | 3.4 (0.5) | 3.5 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response Defined as IGA-C (Investigators Global Assessment) Score ≤ 2 and a SSA-C (Subject Self-Assessment) Score ≤ 2
Description: Composite of Investigators Global Assessment & Subject Self-Assessment on contraction.
  Crow's Feet Wrinkle Scale where severity is scored between 0-4 (0=absent; 4=severe). The same scale is used for the Investigator's Assessment as well as the Subject's Self Assessment. To count, both assessments (on contraction) have to be "responders" defined as Score ≤ 2.
Time Frame: Week 4
Population: Per Protocol (PP) population defined as all treated subjects who had at least one post-baseline visit. No imputation was performed when only incomplete data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | Dose 1 | Dose 2 | Dose 3 | Dose 4
Number analyzed (Participants) | 13 | 8 | 9 | 9 | 8
Participants | 2 | 3 | 4 | 2 | 1

2. Secondary Outcome: Total Number of Observations With a Response Defined as IGA-C Score ≤ 2
Description: Total number of observations with a Score of ≤ 2 on the Investigators Global Assessment on Contraction, IGA-C, using the Crow's Feet Wrinkle Scale, where severity is scored between 0-4 (0=absent; 4=severe). To count, a "responder" is defined as Score ≤ 2. The observation period ranges from the earliest expected onset of action at Week 2 to the likely offset of action by Week 18.
Time Frame: Week 2, 4, 8,12,18
Population: as for outcome 1
Measure: Count of Units; unit: Observations
Units Other Than Participants: Observations
Arm/Group | Vehicle | Dose 1 | Dose 2 | Dose 3 | Dose 4
Number analyzed (Participants) | 13 | 8 | 9 | 9 | 8
Number analyzed (Observations) | 64 | 40 | 45 | 45 | 40
Observations | 16 | 17 | 22 | 16 | 9

3. Secondary Outcome: Total Number of Observations With a Response Defined as SSA-C Score ≤ 2
Description: Total number of observations with a Score of ≤ 2 on the Subject Self-Assessment on Contraction, SSA-C, using the Crow's Feet Wrinkle Scale, where severity is scored between 0-4 (0=absent; 4=severe). To count, a "responder" is defined as Score ≤ 2. The observation period ranges from the earliest expected onset of action at Week 2 to the likely offset of action by Week 18.
Time Frame: Week 2, 4, 8,12,18
Population: as for outcome 1
Measure: Count of Units; unit: Observations
Units Other Than Participants: Observations
Arm/Group | Vehicle | Dose 1 | Dose 2 | Dose 3 | Dose 4
Number analyzed (Participants) | 13 | 8 | 9 | 9 | 8
Number analyzed (Observations) | 64 | 40 | 45 | 45 | 40
Observations | 20 | 19 | 26 | 15 | 8

ADVERSE EVENTS:
Time Frame: 26 Weeks
Arm/Group | Vehicle | Dose 1 | Dose 2 | Dose 3 | Dose 4
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/9 | 0/9 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/9 | 0/9 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/13 | 0/9 | 1/9 | 0/9 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=13) | Dose 1 (N=9) | Dose 2 (N=9) | Dose 3 (N=9) | Dose 4 (N=8)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — PRIOR MYOCARDIAL INFARCTION NOTED ON ECG PRIOR TO STUDY DRUG ADMINISTRATION. CONFIRMED AT WEEK 2 ECG.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study Results are considered Confidential Information that may not be published or disclosed without Sponsor's written consent for a period of five (5) years after completion of the Study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT03326856/Prot_SAP_000.pdf